CLINICAL TRIAL: NCT01628705
Title: Moderated-fat Diet Complemented With Green Tea Reduces oxLDL and Fat Mass in Obese Women: A Randomized, Controlled Clinical Trial
Brief Title: Moderated-fat Diet Complemented With Green Tea Reduces oxLDL and Fat Mass in Obese Women
Acronym: GTRoxLDL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-10808
Record Dates: First submitted 2012-05-17; First posted 2012-06-27 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Nutritional and Metabolic Disease
Keywords: Green tea; oxLDL; fat mass
MeSH Terms: conditions — Metabolic Diseases | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional intervention (Sham Comparator): The subjects were undergoing nutritional intervention.
  Interventions: Other: Nutritional intervention
- Nutritional intervention with green tea (Experimental): The subjects were undergoing nutritional intervention complemented with green tea.
  Interventions: Dietary Supplement: Green tea

INTERVENTIONS:
Other: Nutritional intervention — The subjects were undergoing nutritional intervention was reduced by 500 kcal per day of habitual caloric intake.
  The proportion of daily intake of macronutrient in the moderate-fat diet was: 30% fat (saturated fat <7%, monounsaturated 10-15% and polyunsaturated 10%, respectively to total calories), 15% of protein, and 55% of carbohydrates. The dietary cholesterol was less than 200 mg/day, fiber intake was increased to 25 grams per day (50% soluble fiber).
  Arms: Nutritional intervention
Dietary Supplement: Green tea — The patients drank secha green tea. Subjects of the INT group were instructed on how to prepare the green tea infusion. Each cup was prepared using 3g of dried green tea in 300ml of hot water (temperature 80°C)for 4 min. It was drunk fresh and without sugar. The treatment consisted of 2 cup/day of green tea, one in the morning and one at night. The amount of epigallocathechin-3-gallate was 498mg/day.
  Arms: Nutritional intervention with green tea

SUMMARY:
Background: Obesity is a chronic degenerative disease, considered as cardiovascular risk factor, characterized by systemic inflammation and high levels of oxLDL. Clinical studies have suggested that drink green tea could improve these complications.

Objective: Analyze the effect of a moderate-fat diet complemented with green tea on oxLDL, fat mass and TNFa in obese women.

Design: Randomized, controlled clinical trial. Obese women, without other chronic-degenerative disease were divided using a computer-generated random sequence: control group (CON) with n=32, and intervention group (INT) with n=32; and were instructed to consume a moderate-fat diet, and INT group was instructed to complement the diet with green tea. Anthropometric and biochemical measurements were performed, and oxLDL and TNFa s levels were determined by ELISA. All parameters were realized at baseline and in the 1st, 2nd and 3rd months post-intervention. TNFa mRNA expression was determined by real-time RT-PCR (basal and final). The changes on lipid profile, oxLDL, fat mass and TNFalpha expression were reported of the comparison between basal and final time points. The statistical analysis was performed with SPSS software.

DETAILED DESCRIPTION:
The investigators assessed 114 women with the eligibility criteria: obese women older than 18y, in good health, as determined by a medical history questionnaire, and normal results of clinical laboratory tests excluding lipids. Exclusion criteria was: history of cardiovascular, hepatic, gastrointestinal, or renal disease; no alcoholism, no smoking, no exogenous hormone use or other medication; no supplemental vitamin or infusion drinking (tea, coffee); or treatment for weight loss 3 months before the start of the study. A total of 64 female, Mexican obese patients were included. We conducted the trial between April 2007 and December 2007 in Guadalajara, Jalisco, Mexico. All of the studies were conducted at Departamento de Biología Molecular en Medicina, Hospital Civil "Fray Antonio Alcalde". This study was approved by the Ethical Committee for Human Research, Universidad de Guadalajara (registration number 028/10). The procedures were in accordance with this institution's guidelines and written consent was obtained from each study subject.

ELIGIBILITY:
Inclusion Criteria:

* obese women older than 18 years,
* in good health, as determined by a medical history questionnaire, and
* normal results of clinical laboratory tests excluding lipids

Exclusion Criteria:

* history of cardiovascular, hepatic, gastrointestinal, or renal disease;
* no alcoholism, no smoking, no exogenous hormone use or other medication;
* no supplemental vitamin or infusion drinking (tea, coffee); or
* treatment for weight loss 3 months before the start of the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in low density cholesterol | Change from baseline in lipids, fat mass and TNF aplha levels at 3 months.
  Change in low density cholesterol, change in high density cholesterol, change in triglycerides, change in oxLDL and change in fat mass were assessed at the beginning and at each month during 3 months of intervention. Change in TNF alpha levels was assessed at the beginning and after 3 months. The final changes of all the measures were reported of the comparation between basal and after 3 months.

SECONDARY OUTCOMES:
change in high density cholesterol | baseline, 3 months
change in triglycerides | baseline, 3 months
change in oxLDL | baseline, 3 months
change in fat mass | baseline, 3 months
change in TNF alpha levels | baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: ERIKA MARTINEZ-LOPEZ, PhD, Study Director — University of Guadalajara
Locations (1):
- University of Guadalajara, Guadalajara, Jaliscco, Mexico